CLINICAL TRIAL: NCT04459481
Title: Comparison of Two Bending Angles for Nasotracheal Intubation With a Malleable Vedio Stylet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Juhui Liu, Plastic Surgery Hospital, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PSH-2018-13
Record Dates: First submitted 2020-07-02; First posted 2020-07-07 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: Intubation;Difficult

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 70-degree bending angle group (Experimental): intubation with a 70-degree bending angle
  Interventions: Device: bending angle
- 90-degree bending angle group (Experimental): intubation with a 90-degree bending angle
  Interventions: Device: bending angle

INTERVENTIONS:
Device: bending angle — patients in 70-degree bending angle group are intubated with video stylet at 70-degree bending angle patients in 90-degree bending angle group are intubated with video stylet at 90-degree bending angle

SUMMARY:
Video intubating stylet can be safely and effectively used for nasotracheal intubation, but the optimal bending angle is still unknown. In this study, the optimal bending angle will be determined by comparing the intubation time and success rate of nasotracheal intubation with video intubating stylet at two different bending angles.

DETAILED DESCRIPTION:
intubation will be accomplished at 70 bending angle and 90 degrees bending angle in each group. intubation time, success rate, additional manoeuvres and epistaxis will be recorded and compared.

ELIGIBILITY:
Inclusion Criteria:

* Patients require nasotracheal intubation

Exclusion Criteria:

* fixed, or limited, neck movement, obstructive sleep apnoea, bilateral nasal obstruction or patients with an abnormal coagulation status

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 98 (Actual)
Dates: Start 2020-06-04 (Actual); Primary Completion 2020-11-03 (Actual); Study Completion 2020-11-05 (Actual)

PRIMARY OUTCOMES:
Success rate of nasotracheal intubation | Procedure (From the beginning of intubation to the end of intubation)
  The percentage of successful nasotracheal intubation

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoming Deng, MD, Principal Investigator — Chinese Academy of Medical Sciences and Peking Union Medical College
Locations (1):
- ChineseAMS, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Liu J, Xu W, Jin Z, Deng X. Does Increasing the Bend Angle of a Stylet to 90 degrees Increase the Nasotracheal Intubation Success Rate? J Oral Maxillofac Surg. 2024 Feb;82(2):152-158. doi: 10.1016/j.joms.2023.10.005. Epub 2023 Oct 19. PMID 37926429